CLINICAL TRIAL: NCT02724462
Title: Randomized Trial of An Innovative Smartphone Intervention for Smoking Cessation
Brief Title: Trial of An Innovative Smartphone Intervention for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8317; NCI-2018-02662 (Registry Identifier: NCI / CTRP); RG1001191 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA192849 (NIH)
Record Dates: First submitted 2016-03-24; First posted 2016-03-31 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Smoking
Keywords: smoking cessation; app for quitting smoking
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This is the experimental arm of the study. This includes receiving the novel/experimental smartphone smoking cessation app. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: Smartphone-delivered Intervention (SmartQuit)
- Control (Active Comparator): This is the control arm of the study. This includes receiving the standard of care smartphone smoking cessation app. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: : Smartphone-delivered Intervention (Standard of care app)

INTERVENTIONS:
Behavioral: Smartphone-delivered Intervention (SmartQuit) — The experimental arm includes an intervention using a novel smartphone smoking cessation app.
  Arms: Experimental
Behavioral: : Smartphone-delivered Intervention (Standard of care app) — The control intervention uses a standard of care smartphone smoking cessation app.
  Arms: Control

SUMMARY:
The goal of this study is to determine whether the novel smartphone app (SmartQuit) provides higher quit rates than the current standard smoking cessation app.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* smokes at least five cigarettes daily for at least past 12 months
* wants to quit cigarette smoking in the next 30 days
* if concurrently using any other nicotine or tobacco products, wants to quit using them within the next 30 days
* interested in learning skills to quit smoking
* willing to be randomly assigned to either condition
* resides in US
* has at least daily access to their own personal Apple iPhone, Android, or Windows Phone
* knows how to login and download a smartphone application
* willing and able to read in English
* not using other smoking cessation interventions (including apps or our other intervention studies).
* willing to complete all three follow-up surveys
* provide email, phone, and mailing address.

Exclusion Criteria:

* The exclusion criteria are opposite of the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2503 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, Ph.D., Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santiago-Torres M, Mull KE, Sullivan BM, Cupertino AP, Salloum RG, Triplette M, Zvolensky MJ, Bricker JB. Evaluating the Impact of Pharmacotherapy in Augmenting Quit Rates Among Hispanic Adults in an App-Delivered Smoking Cessation Intervention: Secondary Analysis of a Randomized Controlled Trial. JMIR Form Res. 2025 Jan 31;9:e69311. doi: 10.2196/69311. PMID 39889280
- [Derived] Santiago-Torres M, Mull KE, Sullivan BM, Prochaska JJ, Zvolensky MJ, Bricker JB. Can an Acceptance and Commitment Therapy-Based Smartphone App Help Individuals with Mental Health Disorders Quit Smoking? Depress Anxiety. 2024;2024:1055801. doi: 10.1155/2024/1055801. Epub 2024 Jun 21. PMID 39845432
- [Derived] Santiago-Torres M, Mull KE, Sullivan BM, Bricker JB. Use of e-Cigarettes in Cigarette Smoking Cessation: Secondary Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Nov 9;11:e48896. doi: 10.2196/48896. PMID 37943594
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Santiago-Torres M, Mull KE, Sullivan BM, Ferketich AK, Bricker JB. Efficacy of an acceptance and commitment therapy-based smartphone application for helping rural populations quit smoking: Results from the iCanQuit randomized trial. Prev Med. 2022 Apr;157:107008. doi: 10.1016/j.ypmed.2022.107008. Epub 2022 Mar 4. PMID 35257698
- [Derived] Santiago-Torres M, Mull KE, Sullivan BM, Kendzor DE, Bricker JB. Efficacy and utilization of smartphone applications for smoking cessation among low-income adults: Secondary analysis of the iCanQuit randomized trial. Drug Alcohol Depend. 2022 Feb 1;231:109258. doi: 10.1016/j.drugalcdep.2021.109258. Epub 2021 Dec 31. PMID 35026491
- [Derived] Santiago-Torres M, Mull KE, Sullivan BM, Kwon D, Nollen NL, Zvolensky MJ, Bricker JB. Efficacy and utilization of an acceptance and commitment therapy-based smartphone application for smoking cessation among Black adults: secondary analysis of the iCanQuit randomized trial. Addiction. 2022 Mar;117(3):760-771. doi: 10.1111/add.15721. Epub 2021 Dec 9. PMID 34890104
- [Derived] Bricker JB, Levin M, Lappalainen R, Mull K, Sullivan B, Santiago-Torres M. Mechanisms of Smartphone Apps for Cigarette Smoking Cessation: Results of a Serial Mediation Model From the iCanQuit Randomized Trial. JMIR Mhealth Uhealth. 2021 Nov 9;9(11):e32847. doi: 10.2196/32847. PMID 34751662
- [Derived] Bricker JB, Watson NL, Mull KE, Sullivan BM, Heffner JL. Efficacy of Smartphone Applications for Smoking Cessation: A Randomized Clinical Trial. JAMA Intern Med. 2020 Nov 1;180(11):1472-1480. doi: 10.1001/jamainternmed.2020.4055. PMID 32955554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Smokers were recruited from May 27, 2017 to September 28, 2018, nationally via Facebook ads, a survey sampling company, search engine results, and referral from friends and family.
Groups:
- Experimental: Novel/experimental intervention smartphone smoking cessation app iCanQuit.
- Control: Standard of care control smoking cessation app QuitGuide from NCI.
Period: 3 Month Follow-up Survey
Arm/Group | Experimental | Control
Started | 1254 | 1249
Completed | 1043 | 1050
Not Completed | 211 | 199
Not completed — Lost to Follow-up | 171 | 151
Not completed — Excluded as ineligible after randomization | 40 | 48
Period: 6 Month Follow-up Survey
Arm/Group | Experimental | Control
Started | 1254 | 1249
Completed | 1058 | 1078
Not Completed | 196 | 171
Not completed — Lost to Follow-up | 156 | 123
Not completed — Excluded as ineligible after randomization | 40 | 48
Period: 12 Month Follow-up Survey
Arm/Group | Experimental | Control
Started | 1254 | 1249
Completed | 1040 | 1067
Not Completed | 214 | 182
Not completed — Lost to Follow-up | 174 | 134
Not completed — Excluded as ineligible after randomization | 40 | 48

BASELINE CHARACTERISTICS:
Population: Participants not excluded as ineligible after randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 1214 | 1201 | 2415
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.2 (10.8) | 38.3 (11.0) | 38.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 857 | 843 | 1700
  Male | 357 | 358 | 715
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 105 | 210
  Not Hispanic or Latino | 1109 | 1096 | 2205
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 30 | 58
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 234 | 232 | 466
  White | 836 | 830 | 1666
  More than one race | 89 | 84 | 173
  Unknown or Not Reported | 20 | 21 | 41
Smoking level [Count of Participants; unit: Participants]
  21 or more cigarettes per day | 249 | 239 | 488
  20 or fewer cigarettes per day | 965 | 962 | 1927
Education level [Count of Participants; unit: Participants]
  High school or less education | 500 | 495 | 995
  Some college or more education | 714 | 706 | 1420
CESD-20 Depression Screen [Count of Participants; unit: Participants] — Center for Epidemiological Studies Depression 20-item Scale (CESD-20). The range of possible CESD-20 scores is 0-60, with higher values indicating increased symptom severity. Population: Analysis population includes participants who sufficiently completed the CESD-20 items.
  Participants
    number analyzed (Participants) | 1208 | 1197 | 2405
    CESD-20 score greater than 15 | 583 | 583 | 1166
    CESD-20 score less than or equal to 15 | 625 | 614 | 1239

OUTCOME MEASURES:

1. Primary Outcome: 30-day Point Prevalence Abstinence, Complete-case
Description: Percentage of participants reporting no smoking in the past 30 days, 12 months post-treatment. Participants missing follow-up data are excluded for the complete-case analysis. Exact 2-sided CI was based on the observed proportion of participants.
Time Frame: 12 months post randomization
Population: Participants who reported 30-day point prevalence abstinence at 12 months post-treatment and who were not excluded as ineligible after randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 1040 | 1067
Percentage of participants | 28.2 [25.5 to 31.0] | 21.1 [18.7 to 23.7]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.22 to 1.83]

2. Secondary Outcome: 30-day Point Prevalence Abstinence, Missing=Smoking Imputation
Description: Percentage of participants reporting no smoking in the past 30 days, 12 months post-treatment. Participants missing follow-up data are imputed as still smoking. Exact 2-sided CI was based on the observed proportion of participants.
Time Frame: 12 months post randomization
Population: Participants who were not excluded as ineligible after randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 1214 | 1201
Percentage of participants | 24.1 [21.8 to 26.7] | 18.7 [16.6 to 21.1]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = .001, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.14 to 1.71]

ADVERSE EVENTS:
Time Frame: Approximately 31 months, from the opening of the recruitment window to closure of the data collection window.
Description: This is a smartphone-delivered behavioral intervention, so there were no known risks for serious adverse events, other adverse events, or all-cause mortality.
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/1214 | 0/1201
Serious Adverse Events (participants affected / at risk) | 0/1214 | 0/1201
Other Adverse Events (participants affected / at risk) | 0/1214 | 0/1201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT02724462/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT02724462/Prot_SAP_001.pdf